CLINICAL TRIAL: NCT01914068
Title: A Pilot Study to Investigate Improvements in Physical Fitness and Quality of Life Resulting From a 9 Week Structured Responsive Endurance Training Programme (SRETP) Following Neoadjuvant Chemoradiotherapy Prior to Elective Rectal Cancer Surgery
Brief Title: The Effects of a 9 Week Exercise Programme on Fitness and Quality of Life in Rectal Cancer Patients After Chemoradiotherapy and Before Surgery
Acronym: SRETP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: AintreeNHSTrust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PB-PG-0711-25093; PB-PG-0711-25093 (Other Grant/Funding Number: PB-PG-0711-25093)
Record Dates: First submitted 2013-06-07; First posted 2013-08-01 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Rectal Cancer
Keywords: Neoadjuvant chemoradiotherapy (NACRT); Rectal cancer; Physical fitness; Exercise programme; Surgery; Stage III/IV; Locally advanced operable; patients
MeSH Terms: conditions — Rectal Neoplasms | interventions — Hospitals

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No in hospital exercise training and no exercise advice.
- Exercise Intervention (Active Comparator): In hospital exercise training
  Interventions: Other: Supervised exercise in hospital

INTERVENTIONS:
Other: Supervised exercise in hospital
  Arms: Exercise Intervention

SUMMARY:
Patients' ability to tolerate surgery is associated with physical fitness: less fit patients have an increased rate of death and serious complications following major surgery. Combined chemotherapy and radiotherapy (x-rays) prior to rectal cancer surgery is known as neo-adjuvant chemoradiotherapy (NACRT) and is associated with improved cancer removal but adversely affects physical fitness. In Liverpool, the investigators have pre-pilot data showing that NACRT reduces objectively measured physical fitness (measured by cardiopulmonary exercise testing) in patients having surgery. This pre-pilot study investigated the effects of a 6-week structured responsive endurance training programme (SRETP) after NACRT and before cancer surgery. This programme has improved both their fitness and their health related quality of life(HRQL). Now, the investigators are undertaking a randomised controlled trial to compare changes in patient's physical fitness in response to SRETP with a group of patients who will be given exercise advice. The SRETP group will exercise 3 times a week for 9 weeks. The investigators will make objective measurements of physical fitness in both groups. The investigators will monitor patient's perceptions of the training programme, HRQL, daily activity (using an accelerometer), and outcomes after surgery. The investigators believe that, patients in the exercise group will improve their physical fitness prior to surgery, change behaviour towards exercise, improve activity and HRQL following NACRT. These results will contribute to the design of a large, multi-centre trial to determine whether a SRETP increases physical fitness with a reduction in adverse outcome following surgery. The investigators will conduct an adequately powered randomized controlled trial (RCT) comparing a SRETP with 'exercise advice' in 46 rectal cancer patients. Specifically, we will test the following hypotheses and outcomes: PRIMARY HYPOTHESIS A 9-week, structured responsive endurance training programme (SRETP) compared with a control group (no training) will result in a clinically significant difference in physical fitness (2.0ml/kg/min VO2 at LT) post-NACRT prior to surgery.

SECONDARY OUTCOMES

1. A 9-week SRETP compared with a control group (no training) will result in a clinically significant difference in physical fitness (2.0ml/kg/min VO2Peak) in patients who have had NACRT prior to surgery.
2. SRETP following NACRT and prior to cancer surgery will provide psychological health benefits and improve patient's HRQL (assessed by semi-structured interviews and questionnaires -EORTC QLQ-30 and EQ-5D). This will provide vital exploratory information that will inform a future application to deliver a larger appropriately powered RCT exploring the hypothesis that patients with greater pre-operative fitness will encounter lower postoperative morbidity and mortality. Specifically, these exploratory outcomes are:

EXPLORATORY OUTCOMES

1. To investigate whether SRETP following NACRT and prior to surgery is associated with a change in overall physical activity (assessed by the number of steps while active using an accelerometer).
2. To investigate whether there is a change in the day 7 surgical morbidity (using the Post-Operative Morbidity Survey) and mortality.
3. The effect of SRETP on cancer downstaging post-NACRT (Tumour, Node and Metastasis Staging-TNM staging).

ELIGIBILITY:
Inclusion Criteria:

* All patients listed to undergo elective rectal cancer resection and long course neoadjuvant chemoradiotherapy in the two NHS teaching hospitals (Aintree University Hospital NHS Foundation Trust and Southampton University Hospital NHS Foundation Trust)

Exclusion Criteria:

* Unable to consent.
* Under 18 years of age.
* Unable to perform exercise.
* Any contraindications on the American Thoracic Surgery CPET safety guidelines.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in physical fitness measured by CPET (ml/kg/min) | Pre neoadjuvant chemoradiotherpy(NACRT), post NACRT (week 0 of SRETP) and week 9 of SRETP
  Cardiopulmonary exercise tests will be performed at the time points specified

SECONDARY OUTCOMES:
Quality of life | Pre NACRT (baseline), Mid NACRT (during treatment week3 to 6 dependent on local policies), week 3,9 of SRETP
  Health related quality of life questionnaires will be filled out at each specified time point
Physical activity | Pre NACRT(baseline), Mid NACRT(during treatment 3 to 6 weeks dependent on local policies), week3, 9 of SRETP
  Physical activity monitors, like an armband, will be worn at each specified time point for three days at a time

OTHER OUTCOMES:
Day 7 post operative morbidity score | Day 7 post surgery
  This will be measured on day 7 post surgery with POMS (post operative morbidity score)
TNM Staging | Pre NACRT (baseline), week 9 of SRETP and week 14 pre-surgery
  MRI scans will be performed at each time point specified to investigate cancer downstaging

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Jack, MSc, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- SouthamptonNHSTrust, Southampton, United Kingdom

REFERENCES:
- [Derived] Loughney L, West MA, Moyses H, Bates A, Kemp GJ, Hawkins L, Varkonyi-Sepp J, Burke S, Barben CP, Calverley PM, Cox T, Palmer DH, Mythen MG, Grocott MPW, Jack S; Fit4Surgery group. The effects of neoadjuvant chemoradiotherapy and an in-hospital exercise training programme on physical fitness and quality of life in locally advanced rectal cancer patients: a randomised controlled trial (The EMPOWER Trial). Perioper Med (Lond). 2021 Jun 22;10(1):23. doi: 10.1186/s13741-021-00190-8. PMID 34154675
- [Derived] Loughney L, West MA, Kemp GJ, Rossiter HB, Burke SM, Cox T, Barben CP, Mythen MG, Calverley P, Palmer DH, Grocott MP, Jack S. The effects of neoadjuvant chemoradiotherapy and an in-hospital exercise training programme on physical fitness and quality of life in locally advanced rectal cancer patients (The EMPOWER Trial): study protocol for a randomised controlled trial. Trials. 2016 Jan 13;17:24. doi: 10.1186/s13063-015-1149-4. PMID 26762365